CLINICAL TRIAL: NCT05463185
Title: Effects Of Lymphatic Drainage With And Without Soft Tissue Mobilization On Pain Threshold, Shoulder Mobility And Quality Of Life In Patients With Axillary Web Syndrome.
Brief Title: Effects Of Lymphatic Drainage on Axillary Web Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0511
Record Dates: First submitted 2022-04-15; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Axillary Web Syndrome
Keywords: Axillary web syndrome; Manual lymphatic drainage
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stretching exercises (Experimental): Stretching exercise along with manual lymph drainage
  Interventions: Other: Stretching exercises
- soft tissue mobilization (Experimental): soft tissue mobilization along with manual lymph drainage
  Interventions: Other: Soft tissue mobilization

INTERVENTIONS:
Other: Stretching exercises — Stretching exercises along with manual lymphatic drainage
  Arms: stretching exercises
Other: Soft tissue mobilization — Soft tissue mobilization along with manual lymphatic drainage
  Arms: soft tissue mobilization

SUMMARY:
Axillary web syndrome (AWS) is a common condition related to cording in axilla as a result of axillary lymph nodes dissection surgery in breast cancer patients. This condition comprises of 86% population who underwent breast cancer surgery, but this condition is usually under diagnosed. Usually characterized by pain full cording of soft tissue and contractures at axillary region. This study aims to see the effects of manual lymphatic drainage with or without soft tissue mobilization on patients with axillary web syndrome.

It will be a randomized control trial which will be conducted in cancer centers in government sector hospitals. 30 participants will be enrolled by non probability sampling technique through lottery method into two groups, 15 participants in each group. One group will receive manual lymphatic drainage, while other group will receive manual lymphatic drainage in addition to soft tissue mobilization (3-5 treatment sessions per week for 4 weeks). Base line treatment regimen include stretching, range of motion and strengthening exercises. For outcome measures treatment will be assessed on questionnaires including Disabilities of Arm Shoulder and Hand questionnaire (DASH), Numeric Pain Rating scale (NRS), Breast cancer specific QOL questionnaires (EORTC QLQ-C30, EORTC QLQ BR-23), Patient specific Functional Scale (PSFS), Goniometer and Dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with pain over >3 points, 4 weeks after surgery using
* Numeric Pain Rating scale on upper limb.
* With visible and palpable cords in axilla, arm and breast after surgery.

Exclusion Criteria:

* Acute Thrombosis, Musculoskeletal Disorders,Skin
* Problems: Infections, Osteoarthritis, Rheumatoid Arthritis, Rotator Cuff Syndrome, Adhesive Capsulitis,
* Any other Injury, Trauma and
* Any other Surgery.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females having axillary web syndrome
Enrollment: 20 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-05 (Estimated)

PRIMARY OUTCOMES:
DASH | 10 months
  The DASH (Disabilities of the Arm, Shoulder and Hand) Outcome Measure is a 30-item, self-report questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb.
Numeric Pain Rating Scale | 10 months
  What is the numerical rating scale for pain? The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Goniometer. | 10 months
  A goniometer is a device used in physical therapy to measure a joint's range of motion (ROM).
Breast cancer specific QOL | 10 months
  European Organization for Research and Treatment of Cancer QOL Breast Cancer Specific Version (EORTC QLQ-BR23) . It is a 23-item self-administered breast cancer specific questionnaire, usually administered with the EORTC QLQ-C30, designed to measure QOL in the breast cancer population at various stages and with patients with differing treatment modalities. The assessment is comprised of five domains (body image, sexuality, arm symptoms, breast symptoms, and systemic therapy side effects)
Patient Specific Functional Scale | 10 months
  The Patient Specific Functional Scale (PSFS) is a self-reported valid, reliable, and responsive outcome measure for patients with back, neck, knee and upper extremity problems. It has also been shown to have a high test-retest reliability in both generic lower back pain and knee dysfunction issues.
Dynamometer | 10 months
  dynamometer, or "dyno" for short, is a device for measuring force, moment of force (torque), or power.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, Phd, Principal Investigator — Riphah International University
Locations (1):
- Allied Hosptal, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koehler LA, Haddad TC, Hunter DW, Tuttle TM. Axillary web syndrome following breast cancer surgery: symptoms, complications, and management strategies. Breast Cancer (Dove Med Press). 2018 Dec 20;11:13-19. doi: 10.2147/BCTT.S146635. eCollection 2019. PMID 30588087
- [Background] Leduc O, Sichere M, Moreau A, Rigolet J, Tinlot A, Darc S, Wilputte F, Strapart J, Parijs T, Clement A, Snoeck T, Pastouret F, Leduc A. Axillary web syndrome: nature and localization. Lymphology. 2009 Dec;42(4):176-81. PMID 20218085
- [Derived] Meer TA, Noor R, Bashir MS, Ikram M. Comparative effects of lymphatic drainage and soft tissue mobilization on pain threshold, shoulder mobility and quality of life in patients with axillary web syndrome after mastectomy. BMC Womens Health. 2023 Nov 10;23(1):588. doi: 10.1186/s12905-023-02762-w. PMID 37950230